CLINICAL TRIAL: NCT01829464
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Daily Oral Fasiglifam 25 mg and 50 mg Compared to Placebo When Used in Combination With Sitagliptin in Subjects With Type 2 Diabetes
Brief Title: TAK-875 (Fasiglifam) in Combination With Sitagliptin in Adults With Type 2 Diabetes
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to potential concerns about liver safety (See Detailed Description)
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-875_303; U1111-1124-2270 (Registry Identifier: UTN (WHO))
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Results first posted 2016-06-01 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-04

CONDITIONS: Diabetes
Keywords: Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus | interventions — TAK-875

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): TAK-875 placebo-matching tablets, orally, once daily and sitagliptin 100 mg, tablets, orally for up 24 weeks.
  Interventions: Drug: Placebo
- TAK-875 25 mg (Experimental): TAK-875 25 mg, tablets, orally, once daily and sitagliptin 100 mg, tablets, orally for up to 24 weeks
  Interventions: Drug: TAK-875
- TAK-875 50 mg (Experimental): TAK-875 50 mg, tablets, orally, once daily and sitagliptin 100 mg, tablets, orally for up to 24 weeks
  Interventions: Drug: TAK-875

INTERVENTIONS:
Drug: Placebo — TAK-875 placebo-matching tablets
  Arms: Placebo
Drug: TAK-875 — TAK-875 tablets
  Arms: TAK-875 25 mg
Drug: TAK-875 — TAK-875 tablets
  Arms: TAK-875 50 mg

SUMMARY:
The purpose of this study is to evaluate the effect of TAK-875 (fasiglifam) in combination with sitagliptin on glycemic control in adults with type 2 diabetes.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-875 (fasiglifam). Fasiglifam is being tested to treat people who have type 2 diabetes mellitus and are currently taking sitagliptin (with or without metformin). This study will evaluate glycemic control in people who take fasiglifam plus sitagliptin compared with placebo plus sitagliptin.

The study will enroll approximately 390 patients. Participants will be randomly assigned (by chance, like flipping a coin) to one of the three treatment groups-which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need; all participants will be on 100 mg sitagliptin and may or may not be on metformin background treatment):

* fasiglifam 25 mg
* fasiglifam 50 mg
* Placebo (dummy inactive pill) - this is a tablet that looks like the study drug but has no active ingredient All participants will be asked to take one tablet at the same time each day throughout the study.

This multi-centre trial will be conducted in North America and Latin America. The overall time to participate in this study is approximately 38 weeks. Participants will make 15 visits to the clinic.

Due to potential concerns about liver safety, on balance, the benefits of treating patients with fasiglifam (TAK-875) do not outweigh the potential risks.

For this reason, Takeda has decided voluntarily to terminate the development activities for fasiglifam.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. The participant is male or female and aged 18 years or older with a historical diagnosis of T2DM.
4. The participant meets one of the following criteria:

   * The participant has an HbA1c between 7.5% and 10.5%, inclusive and has been taking a stable dose of sitagliptin 100 mg for at least 8 weeks, with or without metformin, prior to the Screening Visit. A participant who is taking metformin must have received a stable daily dose (≥1500 mg or documented maximum tolerated dose [MTD]) for at least 8 weeks before Screening. This participant will enter the 2-week single-blind Placebo Run-In Period according to Study Schedule A, or;
   * The participant has an HbA1c between 7.5% and 10.5%, inclusive and has been taking any other DPP-IV inhibitor (with or without metformin) for at least 8 weeks prior to the Screening Visit. A participant who is taking metformin must have received a stable daily dose (≥1500 mg or documented MTD) for at least 8 weeks before Screening. This participant will enter the 8-week Switching Period according to Study Schedule B. Following this 8-week period, the participant must qualify for all Inclusion/Exclusion Criteria prior to entering the 2-Week Placebo Run-in Period by completing the Week ( 3) procedures including having an HbA1c level between 7.5% and 10.5%.

   Note: An enrollment cap may be applied to ensure no more than approximately 20% of randomized participants are receiving a DPP-IV inhibitor without metformin at baseline.
5. The participant has had no treatment with antidiabetic agents other than DPP-IV inhibitors and metformin within 2 months prior to Screening (Exception: if a participant has received other antidiabetic therapy for ≤7 consecutive days within the 2 months prior to Screening).
6. The participant has a body mass index (BMI) ≤45 kg/m2 at Screening.
7. Participants regularly using other, non-excluded medications must be on a stable dose for at least 4 weeks prior to screening. However, PRN (as needed) use of prescription or over-the-counter medication is allowed at the discretion of the investigator.
8. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to routinely use adequate contraception from signing of the informed consent throughout the duration of the study and for 30 days after the last dose of study drug.
9. The participant is able and willing to monitor glucose with a home glucose monitor and consistently record his or her own blood glucose concentrations and complete participant diaries.

Exclusion Criteria:

1. Has received any investigational compound within 30 days prior to Screening or has received an investigational antidiabetic drug within 3 months prior to Screening.
2. Has been randomized into a previous TAK-875 study.
3. Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, child, or sibling; biological or legally adopted) or may consent under duress.
4. Donated or received any blood products within 12 weeks prior to Screening or is planning to donate blood during the study.
5. Has a hemoglobin ≤12 g/dL (≤120 gm/L) for males and ≤10 g/dL (≤100 gm/L) for females at the Screening Visit.
6. Has a systolic blood pressure ≥160 mm Hg or diastolic pressure ≥95 mm Hg at Screening (If the participant meets this exclusion criteria, the assessment may be repeated once at least 30 minutes after the initial measurement and a decision will be made based on the second measurement).
7. Has history of cancer that has been in remission for <5 years prior to Screening. (Exception: A history of basal cell carcinoma or stage 1 squamous cell carcinoma of the skin is allowed.)
8. Has alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) levels >2.0x the upper limit of normal (ULN) at Screening.
9. Has a total bilirubin level greater than the ULN at Screening. Exception: if a participant has documented Gilbert's Syndrome, they will be allowed with an elevated bilirubin level per the investigator's discretion.
10. Has a serum creatinine ≥1.5 mg/dL (≥133 μmol/L) [males] and ≥1.4 mg/dL (≥124 μmol/L) [females] and/or estimated glomerular filtration rate (GFR) <60 mL/min/1.73m^2 at Screening.
11. Has uncontrolled thyroid disease.
12. Has a history of laser treatment for proliferative diabetic retinopathy within 6 months prior to Screening.
13. Has had gastric banding or gastric bypass surgery within one year prior to Screening.
14. Has a known history of infection with human immunodeficiency virus (HIV), Hepatitis B virus (HBV), or Hepatitis C virus (HCV).
15. Had coronary angioplasty, coronary stent placement, coronary bypass surgery, myocardial infarction, unstable angina pectoris, clinically significant abnormal electrocardiogram (ECG), cerebrovascular accident or transient ischemic attack within 3 months prior to or at Screening.
16. Has a history of pancreatitis.
17. Has a history of hypersensitivity, allergies or has had an anaphylactic reaction(s) to any component of TAK-875 as well as sitagliptin.
18. Has a history of drug abuse (defined as illicit drug use) or a history of alcohol abuse within 2 years prior to Screening.
19. Received excluded medications prior to the Screening Visit or is expected to receive excluded medications.
20. If female, is pregnant (confirmed by laboratory testing, ie, serum/urine human chorionic gonadotropin (hCG), in females of childbearing potential) or lactating or intending to become pregnant before, during, or within 1 month after participating in this study; or intending to donate ova during such time period.
21. Is unable to understand verbal or written English or any other language for which a certified translation of the approved informed consent is available.
22. Has any other physical or psychiatric disease or condition that in the judgment of the investigator may affect life expectancy or may make it difficult to successfully manage and follow the participant according to the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-05; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Takeda
Locations (86):
- United States (82):
  - Birmingham, Alabama
  - Dothan, Alabama
  - Muscle Shoals, Alabama
  - Phoenix, Arizona
  - Anaheim, California
  - El Cajon, California
  - Long Beach, California
  - Modesto, California
  - North Hollywood, California
  - Norwalk, California
  - Pismo Beach, California
  - San Diego, California
  - Vista, California
  - West Hills, California
  - Boca Raton, Florida
  - Boynton Beach, Florida
  - Bradenton, Florida
  - Clearwater, Florida
  - Cocoa, Florida
  - Doral, Florida
  - Miami, Florida
  - North Miami, Florida
  - Pembroke Pines, Florida
  - Port Orange, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Savannah, Georgia
  - Woodstock, Georgia
  - Boise, Idaho
  - Meridian, Idaho
  - Apex Medical Research, MI, Inc, Chicago, Illinois
  - Chicago, Illinois
  - Avon, Indiana
  - Greenfield, Indiana
  - Muncie, Indiana
  - Council Bluffs, Iowa
  - Topeka, Kansas
  - Owensboro, Kentucky
  - Oxon Hill, Maryland
  - Fall River, Massachusetts
  - St Louis, Missouri
  - Washington, Missouri
  - Omaha, Nebraska
  - Nashua, New Hampshire
  - Elizabeth, New Jersey
  - Haddon Heights, New Jersey
  - Albany, New York
  - Rosedale, New York
  - Calabash, North Carolina
  - Charlotte, North Carolina
  - Greensboro, North Carolina
  - Morganton, North Carolina
  - Winston-Salem, North Carolina
  - Dayton, Ohio
  - Maumee, Ohio
  - Norman, Oklahoma
  - Oklahoma City, Oklahoma
  - Feasterville, Pennsylvania
  - Harleysville, Pennsylvania
  - Levittown, Pennsylvania
  - Uniontown, Pennsylvania
  - Fort Mill, South Carolina
  - Greer, South Carolina
  - Spartanburg, South Carolina
  - Crossville, Tennessee
  - Knoxville, Tennessee
  - Carrollton, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Irving, Texas
  - Katy, Texas
  - Lewisville, Texas
  - McKinney, Texas
  - New Braunfels, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Tomball, Texas
  - Salt Lake City, Utah
  - Burke, Virginia
  - Manassas, Virginia
- Argentina (3):
  - Ciudad Autonoma Buenos Aires, Ciudad Autonoma Buenos Aires
  - Salta, Salta Province
  - Rosario, Santa Fe Province
- Lima, Peru

REFERENCES:
- [Derived] Shavadia JS, Sharma A, Gu X, Neaton J, DeLeve L, Holmes D, Home P, Eckel RH, Watkins PB, Granger CB. Determination of fasiglifam-induced liver toxicity: Insights from the data monitoring committee of the fasiglifam clinical trials program. Clin Trials. 2019 Jun;16(3):253-262. doi: 10.1177/1740774519836766. Epub 2019 Mar 18. PMID 30880443

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 49 investigative sites in the United States from 01 April 2013 to 12 March 2014.
Pre-assignment Details: Participants with historical diagnosis of type 2 diabetes who were inadequately controlled while on sitagliptin 100 milligram(mg) (with/without metformin) or on Dipeptidyl peptidase-4 inhibitor other than sitagliptin(with/without metformin) therapy enrolled in 1 of 3, placebo; fasiglifam 25 mg once daily (QD); fasiglifam 50 mg QD treatment groups.
Groups:
- Placebo: Fasiglifam placebo-matching tablets, orally, once daily and sitagliptin 100 mg, tablets, orally, once daily with or without metformin greater than or equal to (>=) 1500 mg, tablets, orally, once daily for up to 24 weeks.
- Fasiglifam 25 mg QD: Fasiglifam 25 mg, tablets, orally, once daily and sitagliptin 100 mg, tablets, orally, once daily with or without metformin >=1500 mg, tablets, orally, once daily for up to 24 weeks.
- Fasiglifam 50 mg QD: Fasiglifam 50 mg, tablets, orally, once daily and sitagliptin 100 mg, tablets, orally, once daily with or without metformin >=1500 mg, tablets, orally, once daily for up to 24 weeks.
Period: Overall Study
Arm/Group | Placebo | Fasiglifam 25 mg QD | Fasiglifam 50 mg QD
Started | 30 | 31 | 29
Completed | 2 | 2 | 3
Not Completed | 28 | 29 | 26
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Study terminated by sponsor | 25 | 28 | 25
Not completed — Lack of Efficacy | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants who received at least 1 dose of double blind study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Fasiglifam 25 mg QD | Fasiglifam 50 mg QD | Total
Number analyzed (Participants) | 30 | 31 | 29 | 90
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.0 (10.45) | 52.4 (11.61) | 55.2 (8.57) | 54.8 (10.38)
Age, Customized [Number; unit: Participants]
  Less than (<) 65 years | 22 | 27 | 24 | 73
  >= 65 years | 8 | 4 | 5 | 17
Sex/Gender, Customized [Number; unit: Participants]
  Female | 14 | 13 | 16 | 43
  Male | 16 | 18 | 13 | 47
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 6 | 11 | 5 | 22
  Not Hispanic or Latino | 24 | 20 | 24 | 68
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 1 | 3 | 1 | 5
  Black or African American | 3 | 1 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  White | 25 | 26 | 26 | 77
  More than 1 race (multiracial) | 0 | 1 | 0 | 1
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 168.3 (9.26) | 169.0 (10.02) | 166.8 (10.76) | 168.0 (9.96)
Body Mass Index [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 34.49 (5.623) | 32.12 (5.664) | 33.10 (4.315) | 33.23 (5.286)
Region of Enrollment [Number; unit: Participants] — Enrollment in the United States is reported.
  Participants | 30 | 31 | 29 | 90
Smoking Classification [Number; unit: Participants]
  Never smoked | 18 | 19 | 22 | 59
  Current smoker | 7 | 5 | 1 | 13
  Ex-smoker | 5 | 7 | 6 | 18
Baseline Glycosylated Hemoglobin (HbA1c) Category [Number; unit: Participants]
  < 8.5 percent (%) | 16 | 16 | 15 | 47
  >= 8.5% | 14 | 15 | 14 | 43
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 9.291 (8.039) | 8.690 (6.180) | 6.406 (4.390) | 8.154 (6.444)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c at Week 24
Description: The change in the value of HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at Week 24 relative to baseline.
Time Frame: Baseline and Week 24
Population: Full analysis set (FAS) included all randomized participants who received at least 1 dose of double blind study medication and who had a baseline and at least 1 post-baseline assessment.
Measure: Mean (Standard Deviation); unit: Percentage of glycosylated haemoglobin
Arm/Group | Placebo | Fasiglifam 25 mg QD | Fasiglifam 50 mg QD
Number analyzed (Participants) | 26 | 31 | 27
Percentage of glycosylated haemoglobin
  Baseline (n= 26, 31, 27) | 8.39 (0.766) | 8.46 (0.932) | 8.52 (0.956)
  Change at Week 24 (n= 2, 4, 2) | 0.25 (0.495) | -0.80 (0.883) | -1.85 (0.495)

2. Secondary Outcome: Percentage of Participants With HbA1c <7%
Time Frame: Week 24
Population: Due to the relatively limited enrollment and follow-up at the time of study termination, the analysis of percentage of participants with HbA1c <7% at Week 24 was not performed.
Arm/Group | Placebo | Fasiglifam 25 mg QD | Fasiglifam 50 mg QD
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24
Description: The change between the fasting plasma glucose values collected at Week 24 relative to baseline.
Time Frame: Baseline and Week 24
Population: FAS included all randomized participants who received at least 1 dose of double blind study medication and who had a baseline and at least 1 post-baseline assessment.
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | Placebo | Fasiglifam 25 mg QD | Fasiglifam 50 mg QD
Number analyzed (Participants) | 29 | 31 | 28
milligram per deciliter (mg/dL)
  Baseline (n= 29, 31, 28) | 193.76 (50.090) | 184.52 (45.126) | 185.96 (53.767)
  Change at Week 24 (n= 2, 2, 2) | 30.50 (55.861) | -31.50 (16.263) | -85.50 (23.335)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 30 days after the last dose of double-blinded study drug.
Description: At each visit, the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | Fasiglifam 25 mg QD | Fasiglifam 50 mg QD
Serious Adverse Events (participants affected / at risk) | 0/30 | 1/31 | 0/29
Other Adverse Events (participants affected / at risk) | 8/30 | 10/31 | 15/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=30) | Fasiglifam 25 mg QD (N=31) | Fasiglifam 50 mg QD (N=29)
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=30) | Fasiglifam 25 mg QD (N=31) | Fasiglifam 50 mg QD (N=29)
Influenza like illness (General disorders) | 0 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 2
Pain (General disorders) | 0 | 1 | 2
Headache (Nervous system disorders) | 0 | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 2
Amylase increased (Investigations) | 2 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 3
Lipase increased (Investigations) | 2 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.